CLINICAL TRIAL: NCT05067985
Title: SARS-CoV-2 PANDEMIC AND FAILED SPINAL ANESTHESIA: A NIGHTMARE
Brief Title: SARS-CoV-2 PANDEMIC AND FAILED SPINAL ANESTHESIA
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: 72300690-799
Record Dates: First submitted 2021-07-07; First posted 2021-10-05 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-05

CONDITIONS: Regional Anesthesia; SARS-CoV2 Infection
Keywords: regional anesthesia failure; regional anesthesia for SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- SARS-CoV-2 pregnant women: After receiving approval from the local ethics committee and permission to use the hospital archives, we included records of spinal anesthesia performed on confirmed SARS- CoV-2 patients in the Ankara City Hospital between April 2020 and February 2021, as well as related data, in our study. Patients who did not have their data gathered, or whose operation took more than 3 hours due to any reason, were excluded from the study
  Interventions: Procedure: covid 19 spinal anesthesia

INTERVENTIONS:
Procedure: covid 19 spinal anesthesia — this group description covers that all the covid 19 pregnant women which we gave spinal anesthesia for cesarean section procedures. The investigators analyzed them retrospectively.

SUMMARY:
The investigators used a retrospective review of 251 SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) positive patients' cesarean section anesthesia to determine the rate of failed spinal anesthesia, management techniques for failed block, and risk factors that contribute to failure in this study.

DETAILED DESCRIPTION:
All anesthesiologists face a challenge when it comes to the anesthesia of patients with coronavirus disease who are going to have a cesarian section. Patients' and healthcare personnel' safety should be prioritized. Non-emergent procedures in patients with respiratory infections, such as COVID-19 (Coronavirus disease 2019), should be postponed and rescheduled once the infection has been treated. However, some emergency treatments, such as cesarian section, cannot be postponed. So, for COVID 19 patients, which method should be used? According to past studies, the risk of maternal death is 16,7 times higher with general anesthesia than with regional anesthesia (1). Furthermore, general anesthesia, which requires aerosol-generating procedures such as ventilating and intubating patients, has a higher risk of respiratory problems during or after surgery than regional anesthesia. Earlier data on pregnant patients during the COVID 19 pandemic showed no difference in COVID 19-related mortality between pregnant and non-pregnant patients, but a recent study found that pregnancy is associated with a 70% greater risk of death. Another important point is that, when compared to those who are not exposed to tracheal intubation, the transfer of acute respiratory infection to a health care professional during tracheal intubation is 6.6 times higher.

For such reasons, the European and American Societies of Regional Anesthesia jointly issued COVID 19 recommendations stating that regional anesthesia should be preferred over general anesthesia whenever possible, and practice recommendations for regional anesthesia during the pandemic have already been published.

In addition, the American Society of Anesthesiologists and the Society for Obstetric Anesthesiology and Perinatology advise doctors to "consider using neuraxial methods rather than general anesthesia for most cesarian deliveries." In many facilities, single-shot spinal anesthesia is the preferred method for cesarian section. It delivers great anesthesia because of its ease of use, rapid onset of sensory and motor blockage, reliability, ease of mastering, and capacity to provide optimal surgical circumstances; it also minimizes the hazards of general anesthetic while enhancing partition satisfaction. In addition, when compared to general anesthesia, the risk of complications such intraoperative bleeding, surgical site infection, and postoperative pain is lower with spinal anesthesia.

In 1899, August Bier proclaimed spinal anesthesia to be a failure, stating, "Experienced professional, correct technique, single puncture, adequate CSF backflow, effective anesthetic agent!" So, why did it fail? -Capriciousness!!" Single shot spinal anesthesia failure may occur when the subarachnoid space is not reached, or analgesia is not sufficient for surgery after injection. The issue is that if anesthesia fails during COVID 19 procedures, we'll need to develop a new approach for supplementing anesthesia and analgesia cautiously, quickly, and meticulously.

Failed spinal anesthesia can be partial or complete. If anesthesia and analgesia are not achieved within ten minutes after successful intrathecal injection, the bupivacaine spinal anesthetic is regarded to have failed. Partial failure was defined as insufficient extent, quality, or duration of pharmacological action for that procedure, while complete failure was described as no sensory or motor blockage.

Failure of spinal anesthesia necessitates extreme caution, judgment, and technique. If surgery has not yet begun, a partial or total failure can be managed by increasing the Trendelenburg position or administering a second spinal anesthetic. However, if the surgery has already begun, it can be managed by changing positions, injecting local anaesthetic in the operation area by the surgeon, administering sedation with oxygen, opioids, benzodiazepines, or ketamine, and then converting the anesthesia to general anesthesia.

The failure rate of spinal anesthesia is widely distributed, according to researches, ranging from 1 to 17 percent. During spinal anesthesia, the Royal College of Anesthetics proposes a failure rate of 3% in emergencies and 1% for elective procedures. The goal of this study was to determine failure rate and solutions for spinal anesthesia in the context of a COVID 19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* we included records of spinal anesthesia performed on confirmed COVID 19 patients in the Ankara City Hospital between April 2020 and February 2021

Exclusion Criteria:

* Patients who did not have their data gathered, or whose operation took more than 3 hours due to any reason, were excluded from the study.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — all the cesarean section patients included for study
Study Population: we included records of spinal anesthesia performed on confirmed COVID 19 patients in the Ankara City Hospital between April 2020 and February 2021
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
The percentage of failed spinal block | Between implementation of spinal anesthesia to the end of the surgery
  the percentage of failed spinal anesthesia among SARS-CoV-2 positive pregnants who underwent cesarean section under spinal anesthesia

SECONDARY OUTCOMES:
reasons of failure of spinal block | between implementation of spinal anesthesia to the end of the surgery
  possible reasons of inadequate spinal block among SARS-CoV-2 positive parturients who underwent cesarean section under spinal anesthesia
management of failed spinal anesthesia | between implementation of spinal anesthesia to the end of the surgery
  anesthesia, sedation methods to manage failed spinal block for SARS-CoV-2 positive parturients who underwent cesarean section under spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Aygün Güler, md, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Aygun Guler, Ankara, Type A Choice Below ..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warren J, Sundaram K, Anis H, Kamath AF, Mont MA, Higuera CA, Piuzzi NS. Spinal Anesthesia Is Associated With Decreased Complications After Total Knee and Hip Arthroplasty. J Am Acad Orthop Surg. 2020 Mar 1;28(5):e213-e221. doi: 10.5435/JAAOS-D-19-00156. PMID 31478916
- [Background] Neuman MD, Silber JH, Elkassabany NM, Ludwig JM, Fleisher LA. Comparative effectiveness of regional versus general anesthesia for hip fracture surgery in adults. Anesthesiology. 2012 Jul;117(1):72-92. doi: 10.1097/ALN.0b013e3182545e7c. PMID 22713634
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Zambrano LD, Ellington S, Strid P, Galang RR, Oduyebo T, Tong VT, Woodworth KR, Nahabedian JF 3rd, Azziz-Baumgartner E, Gilboa SM, Meaney-Delman D; CDC COVID-19 Response Pregnancy and Infant Linked Outcomes Team. Update: Characteristics of Symptomatic Women of Reproductive Age with Laboratory-Confirmed SARS-CoV-2 Infection by Pregnancy Status - United States, January 22-October 3, 2020. MMWR Morb Mortal Wkly Rep. 2020 Nov 6;69(44):1641-1647. doi: 10.15585/mmwr.mm6944e3. PMID 33151921
- [Background] Tran K, Cimon K, Severn M, Pessoa-Silva CL, Conly J. Aerosol generating procedures and risk of transmission of acute respiratory infections to healthcare workers: a systematic review. PLoS One. 2012;7(4):e35797. doi: 10.1371/journal.pone.0035797. Epub 2012 Apr 26. PMID 22563403
- [Background] Cobb BT, Lane-Fall MB, Month RC, Onuoha OC, Srinivas SK, Neuman MD. Anesthesiologist Specialization and Use of General Anesthesia for Cesarean Delivery. Anesthesiology. 2019 Feb;130(2):237-246. doi: 10.1097/ALN.0000000000002534. PMID 30601216
- [Background] Sng BL, Lim Y, Sia AT. An observational prospective cohort study of incidence and characteristics of failed spinal anaesthesia for caesarean section. Int J Obstet Anesth. 2009 Jul;18(3):237-41. doi: 10.1016/j.ijoa.2009.01.010. Epub 2009 May 17. PMID 19450971
- [Background] Shrestha AB, Shrestha CK, Sharma KR, Neupane B. Failure of subarachnoid block in caesarean section. Nepal Med Coll J. 2009 Mar;11(1):50-1. PMID 19769239
- [Background] Levy JH, Islas JA, Ghia JN, Turnbull C. A retrospective study of the incidence and causes of failed spinal anesthetics in a university hospital. Anesth Analg. 1985 Jul;64(7):705-10. PMID 4014732
- [Background] Fuzier R, Bataille B, Fuzier V, Richez AS, Magues JP, Choquet O, Montastruc JL, Lapeyre-Mestre M. Spinal anesthesia failure after local anesthetic injection into cerebrospinal fluid: a multicenter prospective analysis of its incidence and related risk factors in 1214 patients. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):322-6. doi: 10.1097/AAP.0b013e318217a68e. PMID 21701265
- [Background] van Dillen J, Diesch M, Schutte J, Zwart J, Wolterbeek R, van Roosmalen J. Comparing grades of urgency for classification of cesarean delivery. Int J Gynaecol Obstet. 2009 Oct;107(1):16-8. doi: 10.1016/j.ijgo.2009.05.001. Epub 2009 May 27. PMID 19477442
- [Background] Lucas DN, Yentis SM, Kinsella SM, Holdcroft A, May AE, Wee M, Robinson PN. Urgency of caesarean section: a new classification. J R Soc Med. 2000 Jul;93(7):346-50. doi: 10.1177/014107680009300703. PMID 10928020
- [Background] Kinsella SM. A prospective audit of regional anaesthesia failure in 5080 Caesarean sections. Anaesthesia. 2008 Aug;63(8):822-32. doi: 10.1111/j.1365-2044.2008.05499.x. Epub 2008 Jun 28. PMID 18547291
- [Background] Rukewe A, Adebayo OK, Fatiregun AA. Failed Obstetric Spinal Anesthesia in a Nigerian Teaching Hospital: Incidence and Risk Factors. Anesth Analg. 2015 Nov;121(5):1301-5. doi: 10.1213/ANE.0000000000000868. PMID 26218861
- [Background] Garry M, Davies S. Failure of regional blockade for caesarean section. Int J Obstet Anesth. 2002 Jan;11(1):9-12. doi: 10.1054/ijoa.2001.0903. PMID 15321571
- [Background] Wu J, Chen X, Yao S, Liu R. Anxiety persists after recovery from acquired COVID-19 in anaesthesiologists. J Clin Anesth. 2020 Dec;67:109984. doi: 10.1016/j.jclinane.2020.109984. Epub 2020 Jul 7. No abstract available. PMID 32659378
- [Background] Agarwal A, Agarwal S, Motiani P. Difficulties Encountered While Using PPE Kits and How to Overcome Them: An Indian Perspective. Cureus. 2020 Nov 23;12(11):e11652. doi: 10.7759/cureus.11652. PMID 33251079
- [Background] Adesope OA, Einhorn LM, Olufolabi AJ, Cooter M, Habib AS. The impact of gestational age and fetal weight on the risk of failure of spinal anesthesia for cesarean delivery. Int J Obstet Anesth. 2016 May;26:8-14. doi: 10.1016/j.ijoa.2016.01.007. Epub 2016 Feb 2. PMID 27020240
- [Background] Sharma SK, Gambling DR, Joshi GP, Sidawi JE, Herrera ER. Comparison of 26-gauge Atraucan and 25-gauge Whitacre needles: insertion characteristics and complications. Can J Anaesth. 1995 Aug;42(8):706-10. doi: 10.1007/BF03012669. PMID 7586110
- [Background] Arevalo-Rodriguez I, Munoz L, Godoy-Casasbuenas N, Ciapponi A, Arevalo JJ, Boogaard S, Roque I Figuls M. Needle gauge and tip designs for preventing post-dural puncture headache (PDPH). Cochrane Database Syst Rev. 2017 Apr 7;4(4):CD010807. doi: 10.1002/14651858.CD010807.pub2. PMID 28388808
- [Background] Drasner K, Rigler ML. Repeat injection after a "failed spinal": at times, a potentially unsafe practice. Anesthesiology. 1991 Oct;75(4):713-4. No abstract available. PMID 1817478
- [Background] Steiner LA, Hauenstein L, Ruppen W, Hampl KF, Seeberger MD. Bupivacaine concentrations in lumbar cerebrospinal fluid in patients with failed spinal anaesthesia. Br J Anaesth. 2009 Jun;102(6):839-44. doi: 10.1093/bja/aep050. Epub 2009 Mar 26. PMID 19329469